CLINICAL TRIAL: NCT04738578
Title: A Comparison of Bowel Preparation for Colonoscopy Between Digestive Physicians and Non-digestive Physicians
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MA-1.0
Record Dates: First submitted 2021-01-18; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2019-12

CONDITIONS: Bowel Preparation
Keywords: Predictive factors; Outpatients; Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Outpatients for colonoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnostic accuracy of colonoscopy depends on the quality of bowel preparation, which is a critical element associated with the diagnostic yield, difficulty, time required, and the completeness of colonoscopy. The non-digestive physicians seemed to have a lower quality of bowel preparation compare to the digestive physicians. Therefore, investigators planned to evaluate the risk factors for suboptimal intestinal preparation in outpatients from the perspective of digestive doctors and non-digestive.

ELIGIBILITY:
Inclusion Criteria:

* All outpatients who have already completed the colonoscopy during December 2019 and October 2020.

Exclusion Criteria:

* Patients with incomplete critical information, primary outcome, and baseline characteristics missing as well as examinations in hospitalized patients were excluded.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients undergoing colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 671 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation | One year
  BBPS score (defined as a BBPS score of 2 or higher in any segment and the total BBPS≥6)

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China